CLINICAL TRIAL: NCT05266404
Title: A Randomized, 2-period, 2-treatment, Single-dose, Crossover Study to Assess the Bioequivalence of the Fixed Dose Combination (FDC) of Dapagliflozin 10 mg and Sitagliptin 100 mg, and Dapagliflozin 10 mg and Sitagliptin 100 mg Administered as Individual Tablets in Healthy Subjects
Brief Title: Phase 1 Bioequivalence Study of Dapagliflozin/Sitagliptin FDC vs Loose Combination of Single Components
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1683C00014; 2021-005104-35 (EudraCT Number)
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers (Intended Indication: Type 2 Diabetes Mellitus)
Keywords: Sodium-glucose co-transporter-2 (SGLT2) inhibitor; Dipeptidyl peptidase 4 (DPP4) inhibitor; fixed dose combination (FDC)
MeSH Terms: interventions — dapagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Test Formulation): Dapagliflozin/Sitagliptin FDC tablet (Experimental): Subjects will receive single dose of dapagliflozin/sitagliptin fixed dose combination (FDC) (test formulation).
  Interventions: Drug: Dapagliflozin/sitagliptin FDC
- Treatment B (Reference Formulation): Dapagliflozin+Sitagliptin (Active Comparator): Subjects will receive single dose of dapagliflozin 10 mg tablet + sitagliptin 100 mg tablet co-administered as individual tablets (reference formulation).
  Interventions: Drug: Sitagliptin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin/sitagliptin FDC — Subjects will receive single dose of Dapagliflozin/sitagliptin FDC orally.
  Arms: Treatment A (Test Formulation): Dapagliflozin/Sitagliptin FDC tablet
Drug: Sitagliptin — Subjects will receive 100 mg single dose of Sitagliptin orally.
  Other Names: JANUVIA™
  Arms: Treatment B (Reference Formulation): Dapagliflozin+Sitagliptin
Drug: Dapagliflozin — Subjects will receive 10 mg single dose of Dapagliflozin orally.
  Other Names: FORXIGA™
  Arms: Treatment B (Reference Formulation): Dapagliflozin+Sitagliptin

SUMMARY:
A Study to Assess the Bioequivalence of the fixed dose combination (FDC) of Dapagliflozin and Sitagliptin, and Dapagliflozin 10 mg and Sitagliptin 100 mg administered as individual tablets in Healthy Subject

DETAILED DESCRIPTION:
This study will be a randomized, open-label, 2-period, 2-treatment, single-dose, crossover study in healthy subjects (males and females), performed at a single study center. The study will assess the bioequivalence between a dapagliflozin/sitagliptin FDC tablet (test formulation) and a free combination of dapagliflozin 10 mg + sitagliptin 100 mg co-administered as individual tablets (reference formulation) in fasted conditions to healthy subjects. The study will also assess the Pharmacokinetics (PK) and safety and tolerability of dapagliflozin 10 mg and sitagliptin 100 mg when co-administered as individual tablets and as an FDC tablet.

The study will comprise:

* A Screening Period of maximum 28 days.
* Two Treatment Periods (Treatment A or B)
* A final Safety Follow-up Visit 7 to 14 days after the last dosing with the Investigational medicinal product (IMP) (Treatment A or B).

There will be a minimum washout period of 7 days and a maximum of 14 days between each treatment period.

All subjects will receive a single dose of the following treatments after an overnight fast of 10 hours:

* Treatment A: 1 × dapagliflozin/sitagliptin FDC tablet (test formulation).
* Treatment B: 1 × dapagliflozin 10 mg tablet + 1 × sitagliptin 100 mg tablet co-administered as individual tablets (reference formulation).

Subjects will be randomized to one of 2 treatment sequences: Treatment A followed by Treatment B or Treatment B followed by Treatment A.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative serum pregnancy test at Screening and negative urine pregnancy test within 24 hours prior to investigational Medicinal product (IMP) administration, and must be of non childbearing potential.

  1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.

     Or, if of childbearing potential:
  3. Must not be nursing (breastfeeding).
  4. If heterosexually active, must agree to consistently use an acceptable method of contraception, to avoid pregnancy from at least 4 weeks prior to the first administration of IMP through 90 days after the last dose of IMP.
* Sexually active fertile male subject with partners of childbearing potential must adhere to the contraception methods during the study and until 90 days after the last dose of IMP.
* Have a BMI between 18.5 and 30 kg/m^2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Current or recent (within 3 months of the first IMP dose) gastrointestinal disease that may impact drug absorption and affect the PK of the IMP. Additionally, any gastrointestinal surgery (eg, partial gastrectomy or pyloroplasty), including cholecystectomy, that may impact drug absorption.
* Any major surgery within 4 months of the first IMP dose.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of Screening.
* Donation of > 400 mL of blood within 8 weeks or donation of plasma (except at Screening) within 4 weeks of the first IMP dose.
* Blood transfusion within 4 weeks of the first IMP dose.
* Inability to tolerate oral medication.
* Inability to tolerate venipuncture or inadequate venous access.
* Recent drug or alcohol abuse.
* Excessive intake of alcohol.
* Excessive intake of caffeine-containing drinks or food.
* Use of tobacco-containing or nicotine-containing products.
* History of impaired glucose metabolism.
* Recent vulvovaginal mycotic infections (within 2 months prior to first IMP dose).
* Any other sound medical, psychiatric, and/or social reason, as determined by the Investigator.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at Screening and/or admission to the Clinical Unit.
* Any clinically significant abnormal findings in vital signs at Screening and/or admission to the Clinical Unit.
* Any clinically significant abnormalities on 12-lead ECG at Screening
* Any positive result on screening for serum hepatitis B surface antigen or anti-hepatitis core antibody, hepatitis C antibody, and HIV antibody.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first IMP dose in this study.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to dapagliflozin and sitagliptin or to any of the excipients.
* Positive screen for drugs of abuse at Screening or on each admission to the Clinical Unit or positive screen for alcohol on each admission to the Clinical Unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first IMP dose.
* Use of any prescription drugs or OTC acid controllers within 4 weeks prior to the first IMP dose. Use of any prescribed or non-prescribed medication including analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins, and minerals during the 2 weeks prior to the first IMP dose or longer if the medication has a long half-life.
* Subjects who have previously received dapagliflozin or sitagliptin.
* Subjects who had a severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated).
* Subjects who had the last dose of the COVID-19 vaccine within 7 days of Screening.
* Recent (within 14 days prior to Screening) exposure to someone who has COVID 19 symptoms or positive test results for COVID-19.
* Recent (within 14 days prior to Screening) visit to a healthcare facility where patients with COVID-19 are being treated.
* Subjects who are regularly exposed to COVID-19 as part of their daily life (eg, health care professionals working in COVID-19 wards or at emergency departments).
* Subjects who have positive test results for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) via reverse transcriptase polymerase chain reaction (RT-PCR) before randomization.
* Subject has clinical signs and symptoms consistent with COVID-19 infection or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* Involvement of any AstraZeneca, Parexel, or study site employee or their close relatives.
* Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (ie, during Screening) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who cannot communicate reliably with the Investigator.
* Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from zero to infinity (AUCinf) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.
Maximum observed plasma (peak) drug concentration (Cmax) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRTinf) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.
Terminal rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve (λz) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.
Volume of distribution (apparent) following extravascular administration (based on terminal phase) (Vz/F) | Day 1, Day 2, Day 3 and Day 4
  To demonstrate the fasted-state bioequivalence between a dapagliflozin/sitagliptin FDC tablet relative to dapagliflozin 10 mg + sitagliptin 100 mg when co administered as individual tablets in healthy subjects.

SECONDARY OUTCOMES:
Area under plasma concentration-time curve from zero to infinity (AUCinf) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Maximum observed plasma (peak) drug concentration (Cmax) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRTinf) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Terminal rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve (λz) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Volume of distribution (apparent) following extravascular administration (based on terminal phase) (Vz/F) | Day 1, Day 2, Day 3 and Day 4
  To characterize the PK profiles of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects in a fasted state.
Number of subjects with adverse events (AEs) | From screening (Day -28) to Safety Follow-up (7 to 14 days after the last dosing with the IMP) [up to 66 days]
  To assess the safety and tolerability of single doses of a dapagliflozin/sitagliptin FDC tablet and dapagliflozin 10 mg + sitagliptin 100 mg when co-administered as individual tablets in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Lukka PB, Tang W, Hammarstedt A, Conrad T, Heijer M, Karlsson C, Boulton DW. Racial Comparison of the Pharmacokinetics and Safety of Fixed-dose Combination of Dapagliflozin/Sitagliptin in Western and Korean Healthy Adults. Clin Ther. 2024 Sep;46(9):717-725. doi: 10.1016/j.clinthera.2024.07.007. Epub 2024 Aug 23. PMID 39179458